CLINICAL TRIAL: NCT01322958
Title: Sonographic Assessment and Visualization of Ectopics in Emergency Medicine (SAVE'EM)
Brief Title: Sonographic Assessment and Visualization of Ectopics in Emergency Medicine
Acronym: SAVE'EM
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SAVE'EM
Record Dates: First submitted 2010-04-20; First posted 2011-03-25 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Ectopic Pregnancy
Keywords: bedside ultrasound
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- At Risk of Ectopic Pregnancy: Women who present to the emergency department at UCSF who are at risk of ectopic pregnancy.
  Interventions: Device: Pelvic Ultrasound

INTERVENTIONS:
Device: Pelvic Ultrasound — Pelvic ultrasound performed by the emergency physician
  Other Names: Pelvic Sonogram

SUMMARY:
Observational study of the use of ultrasound by emergency physicians in the evaluation of patients at risk of ectopic pregnancy.

DETAILED DESCRIPTION:
Emergency Physicians who have undergone training according to the American College of Emergency Physicians Guidelines will be evaluated in the accuracy of performing pelvic ultrasounds among patients at risk for ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant females in 1st trimester
* present to emergency department
* complaint of abdominal/pelvic pain or vaginal bleeding

Exclusion Criteria:

* previous ultrasound diagnostic of location of pregnancy

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: women at risk of ectopic pregnancy in emergency department
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2007-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical outcome of the pregnancy | 8 weeks
  To measure the outcome of the study, we will base our results on Sensitivity and Specificity.
  Sensitivity which relates to the number of positive results defined as no intrauterine pregnancies, ectopic pregnancy compared to the Radiologic Gold standard ultrasound which provides us 100% sensitivity. The goal is to reach a sensitivity of (>95%) by our ED physicians.
  Specificity which will be defined as the number of negative studies identified as intrauterine pregnancies compared to the results of the Gold standard radiology ultrasound and by telephone follow up.

CONTACTS AND LOCATIONS:
Overall Officials: John C. Stein, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States